CLINICAL TRIAL: NCT04401553
Title: First Tier Versus Second Tier Antibiotics for Surgical Site Infections Following Hysterectomy In the Patients With a Beta-Lactam Allergy: A Prospective, Randomized, Single-Blinded Clinical Trial
Brief Title: Prophylactic Antibiotics for Surgical Site Infections and Beta-Lactam Allergy
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The study never initiated.
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Mark Haney, Assistant Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: STU-2020-0317
Record Dates: First submitted 2020-05-20; First posted 2020-05-26 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Surgical Site Infection; Beta-lactam Allergy
MeSH Terms: conditions — Surgical Wound Infection | interventions — Cephalosporins; Vancomycin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- First Tier Antibiotic (Experimental): First tier antibiotics, cephalosporin, will be given before anesthesia induction in the subjects with a history of allergy-like event to beta-lactam
  Interventions: Drug: cephalosporin
- Second Tier Antibiotic (Active Comparator): Second tier antibiotics, vancomycin, will be given before anesthesia induction for infection prevention in the subjects with a history of allergy-like event to beta-lactam
  Interventions: Drug: Second tier antibiotic (Vancomycin)

INTERVENTIONS:
Drug: cephalosporin — First tier antibiotics, cephalosporin, will be given before anesthesia induction in the subjects with a history of allergy-like event to beta-lactam
  Arms: First Tier Antibiotic
Drug: Second tier antibiotic (Vancomycin) — Second tier antibiotics, vancomycin, will be given before anesthesia induction for infection prevention in the subjects with a history of allergy-like event to beta-lactam (standard of care)
  Other Names: Vancomycin
  Arms: Second Tier Antibiotic

SUMMARY:
Postoperative surgical site infection (SSI) is associated with unnecessary use of heath care resources including prolonged hospitalization and increased hospital readmission. Perioperative antibiotic prophylaxis is one of the most important strategies for prevention of SSI. If there is a beta-lactam allergy, second tier antibiotics (vancomycin and clindamycin) are recommended alternatives to first- and second-generation cephalosporins because of fears of possible allergy.

This prospective, randomized, and single-blinded clinical trial is designed to examine causality between second tier antibiotics use and surgical site infections in the subjects with a documented unverified penicillin allergy. Unverified beta-lactam allergy could be associated with antimicrobial treatment failure with second tires antibiotics during postoperative period.

DETAILED DESCRIPTION:
In this prospective, randomized, single-blinded clinical trial, eligible subjects will be identified based on scheduled elective hysterectomy. Subjects with documented beta-lactam allergy in their chart will be evaluated to differentiate true allergy and allergy-like events. Subjects with history of allergy-like event to beta-lactam antibiotics will be randomized to either receive first tier antibiotic or second tier antibiotics before anesthesia induction.

Preoperative Screening of Allergy The potential subjects' history of allergy will be reviewed according to described criteria of allergy like events. Subjects with documented anaphylaxis to first tier and second tier antibiotics will be excluded. Only subjects with a history of previous allergic-like event after beta-lactam antibiotic will be enrolled to the study.

An allergy self-screening questionnaires will be reviewed before the surgery to identify true allergy or allergy-like event to beta-lactam (penicillin). Allergic-like events include nausea, vomiting, feeling dizziness, dermatitis seen after beta-lactam antibiotic, or any other description of hypersensitivity reactions other than anaphylactic shock, angioedema, laryngeal spasm, and shock. Administration of the potential confounding drugs such as antihistamines, systemic and topical corticosteroids and potential confounding diagnosis such as autoimmune disease will be also reviewed together with allergy history of the subjects to differentiate true hypersensitivity and allergy-like events to penicillin and other beta-lactam antibiotics.

Postoperative Follow-up for SSI:

Subjects will be followed postoperatively for post-discharge SSIs or clostridium infection by reviewing medical records and contacting via phone and survey. If the subject received care outside the clinic, their provider will be contacted to obtain outside clinic record with subject permission.

The post-discharge SSIs will be followed according to the SSI surveillance survey protocol (Harrington et al. 2013). A combination of methods listed below will be used to detect post-discharge SSI.

1. Identification of subject readmitted with SSI (medical record review)
2. Detection of SSI at outpatient clinic, other return visit to hospital or review by healthcare staff (direct observation of the wound by health professional)
3. Telephone interviews or questionnaire (self-reported SSI)

   * Early post-operative follow-up (30-days) Subjects will be contacted via phone at 30 days (±3 days) post-operatively to determine if they have been told by a physician they have a wound infection or if their post-operative antibiotics will extend due to concern for wound infection.
   * Late post-operative follow-up (90-days) A redcap survey will be sent at postoperative 90 days to review any possible wound infection.

Surgical Site infection (Wound) Classification Based on standard definitions from the US Centers for Disease Control and Prevention for SSI, the wound infections will be classified as

1. superficial incisional (infection occurred within 30 days after any operative procedure and involved only skin and subcutaneous tissue of the incision),
2. deep incisional primary/secondary (infection occurred within 31-90 days after the operative procedure and involved deep soft tissues of the incision), or organ/space (infection occurred within 31-90 days after the operative procedure and involved any part of the body deeper than the fascia/muscle layers that was opened or manipulated during the operative procedure.

Criteria of the SSI decision for the female reproductive tract infection (excluding endometritis or vaginal cuff infections) must meet at least one of the following criteria:

* Criterion 1: Organisms are cultured from tissue or fluid from affected site.
* Criterion 2: There is an abscess or other evidence of infection of affected site seen during a surgical operation or histopathological examination.
* Criterion 3: The subjects have two of the following signs or symptoms with no other recognized cause: fever (>38°C), nausea, vomiting, pain, tenderness, or dysuria, and at least one of the following: (a) organisms cultured from blood (b) diagnosis by physician.

The SSI criteria listed above will be applied to the self-reported SSI. Type of SSI will not be recorded in self-reported SSI. Wound type will be decided according to documentation of clinician who evaluates the wound. If a superficial SSI progresses into a deep SSI, it will be reported as the deep SSI only. It may be possible for a subject to have an organ/space SSI in addition to a SSI affecting the incision (superficial or deep) but if more than one SSI is reported each must meet the case definition.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects age 18 and older
2. Subjects undergoing open total abdominal hysterectomy
3. Subjects with documented beta-lactam allergy

Exclusion Criteria:

1. Subjects with documented anaphylaxis to Tier 1 or Tier 2 antibiotics
2. Surgical procedure within 30 days prior to hysterectomy
3. Robotic hysterectomy
4. Presence of multidrug resistant organism such as methicillin-resistant Staphylococcus aureus (MRSA)
5. Immunocompromised subject
6. Cognitive deficits 7- Chronic Kidney Disease or patients on dialysis 8- Severe liver disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-08-16 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Surgical site infections during early postoperative period | Early post-operative period within a 30-day after hysterectomy
  Incidence of surgical site infections after hysterectomy

SECONDARY OUTCOMES:
Infectious hospital readmission | the postoperative period within a 90-days after hysterectomy
  Incidence of infectious hospital readmission

CONTACTS AND LOCATIONS:
Overall Officials: Mark Haney, MD, Study Director — University of Texas Southwestern Medical Center